CLINICAL TRIAL: NCT01645761
Title: Additive Effect of Endonase on Eradication Rate of the 7-day Standard Proton Pump Inhibitor-based Triple Therapy for Helicobacter Pylori
Brief Title: Additive Effect of Endonase on Eradication Rate of First Line Therapy for Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Yeonsoo Kim, Assistant Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSHH Endonase 1; CLDD 1 (Other: CSHH CLDD 1)
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Gastric Ulcer Associated With Helicobacter Pylori
Keywords: Helicobacter pylori eradication; Peptic ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPI-based triple therapy with endonase (Experimental): 7-day standard proton pump inhibitor-based triple therapy (the standard dosage of PPI, 1,000 mg of amoxicillin and 500 mg of clindamycin twice daily for one week) plus 20,000 units of endonase twice daily for one week.
  Interventions: Drug: Endonase
- PPI-based triple therapy (No Intervention): 7-day standard proton pump inhibitor-based triple therapy (the standard dosage of PPI, 1,000 mg of amoxicillin and 500 mg of clindamycin twice daily for one week)

INTERVENTIONS:
Drug: Endonase — PPI- based triple therapy with endonase
  Arms: PPI-based triple therapy with endonase

SUMMARY:
Endonase, a kind of protease, is known to cause both extensive degradation of mucins and a reduction in mucus viscosity. As part of the search for more effective forms of therapy against H. pylori when it colonizes not only the surface of the surface mucosal cells but also the surface mucous gel layer covering the mucosal surface of the stomach. The investigators decided to investigate whether or not endonase might have additive effect of pronase on the efficacy of eradication therapy against Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

Male or Female with 18 years or more of age without history of H. pylori eradication AND

1. Patients with H. pylori associated peptic ulcer in scar stage, OR
2. Non-ulcer dyspepsia patients with H. pylori infection

Exclusion Criteria:

1. Under 18 years, OR
2. Patients with a history of previous treatment of H. pylori infection, OR
3. Pregnant or Breast feeding women, OR
4. Patients with severe renal, liver, or heart disease, OR
5. Patients with gastric malignancy, OR
6. Patients with a history of drug allergy or hypersensitivity, OR
7. Patients who had received treatment with antibiotics or proton pump inhibitors, H2 Blocker, Bismuth preparation, Anticoagulant, Ketoconazole, Glucocorticoid during the 2 weeks preceding endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Eradication rate | 4 weeks
  Intention-to-treat analysis and per-protocol analysis to compare the eradication rate of the 7-day standard PPI-based triple therapy plus endonase with that of the 7-day standard PPI-based triple therapy

SECONDARY OUTCOMES:
Number of participants with adverse events | 4 weeks
  Difference in the number of participants with adverse events between patients receiving standard triple therapy plus endonase and patients receiving control treatment
Number of participants taking over 85% of medicine | 4 weeks
  Difference in the number of participants taking over 85% of medicine between patients receiving standard triple therapy plus endonase and patients receiving control treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jin Bong Kim, MD, Study Chair — Department of Internal Medicine, Hallym university college of medicine; Yeon Soo Kim, MD, PhD., Study Director — Department of Internal Medicine, Hallym University College of Medicine; Chang Seok Bang, MD, Principal Investigator — Department of Internal Medicine, Hallym University of College of Medicine
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Derived] Bang CS, Kim YS, Park SH, Kim JB, Baik GH, Suk KT, Yoon JH, Kim DJ. Additive Effect of Pronase on the Eradication Rate of First-Line Therapy for Helicobacter pylori Infection. Gut Liver. 2015 May 23;9(3):340-5. doi: 10.5009/gnl13399. PMID 25167799